CLINICAL TRIAL: NCT03091673
Title: A Phase 3 Study to Evaluate the Glucose Response of G-Pen (Glucagon Injection) in Pediatric Patients With Type 1 Diabetes
Brief Title: Glucose Response of G-Pen (Glucagon Injection) in Pediatric T1D Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xeris Pharmaceuticals (Industry)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XSGP-302
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Results first posted 2018-11-16 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- G-Pen (glucagon injection) 0.5 mg (Experimental): A single 0.5 mg subcutaneous (SC) injection of G-Pen (glucagon injection)
  Interventions: Drug: Glucagon
- G-Pen (glucagon injection) 1.0 mg (Experimental): A single 1.0 mg subcutaneous (SC) injection of G-Pen (glucagon injection)
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon — 0.5 or 1.0 mg of pre-mixed liquid Xeris glucagon delivered via auto-injector
  Other Names: G-Pen (glucagon injection)

SUMMARY:
This is a sequential efficacy and safety study in pediatric patients with type 1 diabetes. Subjects will be administered insulin to induce a low normal glycemic state and will then receive an age-appropriate dose of G-Pen (glucagon injection) in a clinical research center (CRC) or comparable setting.

DETAILED DESCRIPTION:
This is an open-label, Phase 3 sequential efficacy and safety study in pediatric patients ages 2-17 with type 1 diabetes. Patients will complete the screening procedures up to 30 days before dosing to determine eligibility before enrollment to the treatment phase.

The procedure to evaluate the efficacy of G-Pen (glucagon injection) consists of inducing a low normal glycemic state by administration of insulin. Subjects ages 2-11 will then be given a 0.5 mg dose of G-Pen, while subjects ages 12-17 will receive a 1 mg dose of G-Pen. Subjects ages 12-17 will return for a second visit 1-4 weeks later and will receive a 0.5 mg dose of G-Pen when in a low normal glycemic stare. Plasma glucose and glucagon levels will be monitored for 90 and 180 minutes post-dosing, respectively, at all visits.

A follow-up phone call as a safety check will be conducted 3 - 14 days following administration of the final dose.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with T1D for at least 6 months at Screening.
* current usage of daily insulin treatment.

Exclusion Criteria:

* pregnant or nursing
* renal insufficiency
* hepatic synthetic insufficiency
* aspartate or alanine aminotransferase > 3 times the upper limit of normal
* hematocrit less than or equal to 30%
* use of > 2.0 U/kg total insulin dose per day
* inadequate venous access
* current seizure disorder
* history of pheochromocytoma or disorder with increased risk of pheochromocytoma
* history of insulinoma
* history of glycogen storage disease.
* active use of alcohol or drugs of abuse
* administration of glucagon within 14 days of the first treatment visit
* participation in other studies involving an investigational drug or device within 30 days

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Women & Children's Hospital of Buffalo, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Dose
Arm/Group | G-Pen (Glucagon Injection) 0.5 mg | G-Pen (Glucagon Injection) 1.0 mg
Started | 31 | 0 (All 31 subjects received the 0.5 mg dose during period 1.)
Completed | 31 | 0
Not Completed | 0 | 0
Period: Second Dose
Arm/Group | G-Pen (Glucagon Injection) 0.5 mg | G-Pen (Glucagon Injection) 1.0 mg
Started | 0 (No subjects received the 0.5 mg dose during period 2.) | 11 (Only the 11 study subjects ages 12-<18 years were assigned the 1 mg dose during period 2.)
Completed | 0 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subjects 2 to <6 Years of Age: Study subjects at least 2, but less than 6 years of age at the time of dosing
- Subjects 6 to <12 Years of Age: Study subjects at least 6, but less than 12 years of age at the time of dosing
- Subjects 12 to <18 Years of Age: Study subjects at least 12, but less than 18 years of age at the time of dosing
- Total: Total of all reporting groups
Arm/Group | Subjects 2 to <6 Years of Age | Subjects 6 to <12 Years of Age | Subjects 12 to <18 Years of Age | Total
Number analyzed (Participants) | 7 | 13 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.96 (1.1) | 9.95 (2.25) | 15.48 (1.58) | 10.79 (4.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 16
  Male | 2 | 8 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 13 | 11 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 5 | 12 | 11 | 28
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 13 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Glucose
Description: The primary endpoint for this study is an evaluation of change in plasma glucose following treatment with G-Pen, with an emphasis on the increase from baseline to 30 minutes post-dosing.
Time Frame: 0-30 minutes
Population: All enrolled subjects.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Subjects 2 to <6 Years of Age: Study subjects at least 2, but less than 6 years of age at the time of receiving a 0.5 mg dose of G-Pen.
- Subjects 6 to <12 Years of Age: Study subjects at least 6, but less than 12 years of age at the time of receiving a 0.5 mg dose of G-Pen.
- Subjects 12 to <18 Years of Age: Study subjects at least 12, but less than 18 years of age at the time of receiving a 1 mg dose of G-Pen.
Arm/Group | Subjects 2 to <6 Years of Age | Subjects 6 to <12 Years of Age | Subjects 12 to <18 Years of Age
Number analyzed (Participants) | 7 | 13 | 11
mg/dL | 81.4 (18.3) | 84.2 (25.3) | 54.0 (27.3)
Statistical Analysis 1: Comparison: Subjects 2 to <6 Years of Age vs Subjects 6 to <12 Years of Age vs Subjects 12 to <18 Years of Age; Test type: Other; p < 0.001, t-test, 2 sided — P-value was computed using a t-test to determine if change in plasma glucose from baseline to 30 minutes was zero

2. Secondary Outcome: Time for Plasma Glucose to Increase by ≥25 mg/dL
Description: Time for plasma glucose to increase by ≥25 mg/dL from baseline will be analyzed descriptively for each age cohort.
Time Frame: 0-90 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Subjects 2 to <6 Years of Age | Subjects 6 to <12 Years of Age | Subjects 12 to <18 Years of Age
Number analyzed (Participants) | 7 | 13 | 11
minutes | 16.4 (3.78) | 16.2 (4.63) | 26.6 (9.51)

3. Secondary Outcome: Plasma Glucagon Area Under the Curve
Description: Plasma glucagon area under the curve (AUC) for each age cohort will be analyzed descriptively.
Time Frame: 0-90 minutes
Measure: Mean (Standard Deviation); unit: min*mg/dL
Arm/Group | Subjects 2 to <6 Years of Age | Subjects 6 to <12 Years of Age | Subjects 12 to <18 Years of Age
Number analyzed (Participants) | 7 | 13 | 11
min*mg/dL | 14440.8 (2114.9) | 14392.3 (2698.4) | 13105.5 (13105.45)

4. Secondary Outcome: Plasma Glucagon Cmax
Description: Plasma glucagon maximum concentration for each age cohort will be analyzed descriptively.
Time Frame: 0-180 minutes
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Subjects 2 to <6 Years of Age | Subjects 6 to <12 Years of Age | Subjects 12 to <18 Years of Age
Number analyzed (Participants) | 7 | 13 | 11
mg/dL | 202.3 (35.9) | 216.3 (51.2) | 199.0 (57.0)

5. Secondary Outcome: Plasma Glucagon Tmax
Description: Plasma glucagon time to maximum concentration for each age cohort will be analyzed descriptively.
Time Frame: 0-180 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Subjects 2 to <6 Years of Age | Subjects 6 to <12 Years of Age | Subjects 12 to <18 Years of Age
Number analyzed (Participants) | 7 | 13 | 11
minutes | 66.6 (10.5) | 68.5 (15.3) | 81.2 (14.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signing of informed consent through the follow-up phone call, which was completed 3-14 days after the last dose of treatment. The maximum adverse event (AE) collection period was 44 days for subjects receiving a single dose, and 72 days for subjects receiving 2 doses of G-Pen.
Arm/Group | Subjects 2 to <6 Years of Age | Subjects 6 to <12 Years of Age | Subjects 12 to <18 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 5/7 | 12/13 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects 2 to <6 Years of Age (N=7) | Subjects 6 to <12 Years of Age (N=13) | Subjects 12 to <18 Years of Age (N=11)
Nausea (Gastrointestinal disorders) | 3 (4) | 7 (7) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03091673/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT03091673/SAP_001.pdf